CLINICAL TRIAL: NCT00385528
Title: Effects of a Multi-Faceted Psychiatric Intervention Targeted at the Complex Medically Ill: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCS-3200-066718
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Rheumatoid Arthritis; Diabetes
Keywords: Case complexity; INTERMED; Consultation liaison psychiatry; depression
MeSH Terms: conditions — Arthritis, Rheumatoid; Diabetes Mellitus; Depression

INTERVENTIONS:
Behavioral: Multi-faceted psychiatric intervention

SUMMARY:
Background: somatic patients with psychiatric co-morbidities are a major challenge for the health care system. This study evaluated a psychiatric intervention targeted at the complex medically ill identified by means of the INTERMED, an instrument to assess case complexity.

Methods: of 885 rheumatology inpatients and diabetes outpatients who were assessed for eligibility, 247 were identified as complex (INTERMED score > 20) and randomized to the intervention (N=125, 84 rheumatology and 41 diabetes patients) or care as usual (N=122, 78 rheumatology and 44 diabetes patients). Intervention consisted of counseling by a psychiatric nurse, referral to a liaison psychiatrist, or a multidisciplinary case conference. Baseline and follow up at months 3, 6, 9 and 12 measured prevalence of major depression (MINI), depressive symptoms (CES-D), physical and mental health (SF-36), quality of life (EuroQol), hospitalizations (rheumatology patients) and HbA1c levels (diabetic patients).

DETAILED DESCRIPTION:
Of the 885 that assessed for eligibility (see Figure 2), 184 (20.8%) met exclusion criteria, such as not speaking French (N=43), severe cognitive disturbances (N=27) or hospitalization for less than 3 days (N=28); 6.2% refused to participate (N=55). Of the remaining patients (N= 701), 64.8% (N=454) did not qualify as complex patients (INTERMED score < 20). The remaining 247 patients were randomized, 125 (84 rheumatology inpatients and 41 diabetes outpatients) to the intervention and 122 to care as usual (78 rheumatology inpatients and 44 diabetes outpatients). With regard to sociodemographics and baseline measurements (including the above mentioned strata of the rheumatology patients and the different types of diabetes), intervention and care as usual group did not differ at baseline (see Table 1). More than half of the sample (61% of the intervention group and 56% of the care as usual group) suffered from major depression.

In the intervention arm, most patients (N = 107) received an intervention conducted by the psychiatric liaison nurse; the interventions, effectuated as single interventions or combined, consisted of "facilitating emotional expression" (73%), "giving practical advice" (71%), "promoting life narrative" (48%) and "providing psycho-educational interventions" (44%). For about half of the patients in the intervention group (N = 76) also other types of interventions were proposed, such as referral to a liaison psychiatrist (N = 36), psychiatric advice to the treating physician (N = 32) or interdisciplinary case conferences (N = 8). A minority of patients (N=13) did not receive any treatment (due to no indication for a psycho-social intervention or patients lacking motivation) (N=13). The liaison nurses, who effectuated the intervention and organized psychiatric referral, psychiatric advice to the treating physician and interdisciplinary case conferences, were supervised weekly for an hour by a senior psychiatrist (FS) or an experienced psychiatric liaison nurse (YD).

Between 62% and 70% of the patients of the intervention arm and between 57% to 69% of patients of the usual care arm provided complete follow up data at the four time points (see Figure 2). Patients with missing data did not differ from patients with complete data with regard to age, sex, educational and professional status, baseline quality of life and depression on each of the four follow up assessments.

Effects of intervention

In Table 2 and Figures 3-7, comparisons between patients in the intervention arm on and usual care arm on the main outcomes are presented. Overall, the intervention was associated with less depression and higher levels of quality of life during follow up. Using statistical tests to evaluate differences at each of the separate follow up points, statistically significant differences are observed with regard to the prevalence of major depression at 12 months, physical health at 3 months and quality of life at 3, 6, and 12 months (see Table 2).

ELIGIBILITY:
Inclusion Criteria:

* PAtients between 19-65 years old,
* inpatient rheumatology patients and diabetes outpatients,
* case complexity above 21 on the INTERMED

Exclusion Criteria:

* cognitive failure,
* not french speaking,
* terminal illness

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Psychological distress, quality of life

SECONDARY OUTCOMES:
health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich C Stiefel, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University Hospital Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] de Jonge P, Huyse FJ, Slaets JP, Sollner W, Stiefel FC. Operationalization of biopsychosocial case complexity in general health care: the INTERMED project. Aust N Z J Psychiatry. 2005 Sep;39(9):795-9. doi: 10.1080/j.1440-1614.2005.01684.x. PMID 16168037